CLINICAL TRIAL: NCT02364115
Title: Randomized Controlled Trial Comparing Conventional Radiotherapy With Stereotactic Body Radiotherapy in Patients With Bone Metastases - VERTICAL Study
Brief Title: Randomized Trial Comparing Conventional Radiotherapy With Stereotactic Radiotherapy in Patients With Bone Metastases - VERTICAL Study
Acronym: VERTICAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Prof. dr., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL49316.041.14
Record Dates: First submitted 2015-02-01; First posted 2015-02-16 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Spinal Metastases; Bone Metastases
Keywords: Spinal metastases; Spinal metastatic disease; Stereotactic Body Radiotherapy; Response; Bone metastases
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stereotactic Body Radiotherapy (Experimental): MRI-based, cone beam CT-guided SBRT delivery of a single dose of 18 Gray (Gy) on the visible metastasis, and 8 Gy on the bony compartment containing the metastasis (e.g. the affected vertebra or pedicle).
  Interventions: Radiation: Stereotactic Body Radiotherapy
- Conventional Radiotherapy (No Intervention): Delivery of a single fraction of 8 Gy using virtual simulation

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy
  Other Names: Stereotactic Radiosurgery
  Arms: Stereotactic Body Radiotherapy

SUMMARY:
The purpose of the study is to investigate effectiveness of stereotactic body radiotherapy in patients with bone metastatic disease.

DETAILED DESCRIPTION:
Rationale: Bone metastases are a frequent distant manifestation of solid tumours, and many bone metastases are located in the spine. These patients mostly present with severe (back) pain which reduces quality of life. The primary treatment for pain management is a single-fraction low dose external beam radiation therapy (EBRT), effective in achieving pain reduction in around 60% of patients, of whom 0-23% experience complete pain response. Recently, there is growing evidence that Stereotactic Body Radiotherapy (SBRT) achieves a much higher pain response due to the higher dose administered. In retrospective and a few prospective case series, SBRT for spinal, and also non-spinal metastases has been demonstrated to be safe, and efficacious. However, no randomized controlled trials have been performed.

Objective: To study whether the pain response after three months in patients with osseous metastatic disease increases after SBRT in comparison to low dose EBRT.

Study design: Randomized controlled trial, the VERTICAL study, nested within the PRESENT cohort.

Study population: Eligible patients are MRI-compatible patients with radiographic evidence of bone metastases at the radiotherapy department. Fifty-five patients are recruited in both control and intervention arm.

Intervention: Patients will undergo MRI-based, cone beam CT-guided SBRT and will receive a single dose of 18 Gray (Gy) on the visible metastasis, and 8 Gy on the bony compartment containing the metastasis (e.g. the affected vertebra or pedicle).

Main study parameters/endpoints: The primary endpoint is pain control at three months after radiotherapy. Secondary outcomes are, among others, the occurrence of vertebral compression fracture (VCF) and radiation-induced myelopathy, local tumour control and evaluation of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of bone metastases
* For spinal lesions; per lesion no more than 3 consecutive spine segments involved with one unaffected vertebral body above and below
* No more than 2 painful lesions needing treatment
* Histologic proof of malignancy
* No compression of spinal cord
* No or mild neurological signs (i.e. radiculopathy, dermatomal sensory change, and muscle strength of involved extremity is Medical Research Council (MRC) 4/5
* Medically inoperable or patient refused surgery
* Karnofsky performance score (KPS) > 50
* Numeric rating scale (NRS) > 3
* Age > 18 years
* Written informed consent
* Filling out PRESENT-questionnaires

Exclusion Criteria:

* Lesion in C1 or C2
* Radio-sensitive histology such as multiple myeloma, lymphoma, small cell, germ cell
* Spinal MRI cannot be completed for any reason (in according with the MRI protocol of the Department of Radiology)
* Impossible to delineate metastasis and organs at risk (OAR) due to artifacts on CT or MRI from previous surgical stabilization
* Unable to undergo SBRT treatment, according to treating doctor's opinion
* Epidural disease
* Severe, worsening or progressive neurological deficit
* Unstable lesion requiring surgical stabilization
* Patient with < 3 months life expectancy
* Previous EBRT or SBRT to same level
* Chemotherapy or systemic radionuclide delivery within 24 hours before and after SBRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Complete or partial pain response after radiation, defined according to the International Bone Metastases Consensus Endpoints for Clinical Trials. | 3 months
  The primary endpoint of this study is complete or partial pain response after SBRT or EBRT after three months. Complete and partial response, but also possible pain progression or indeterminate response, will be defined according to the International Bone Metastases Consensus Endpoints for Clinical Trials.

SECONDARY OUTCOMES:
Health-Related Quality of Life | at 2, 4, 6, 8 weeks, 3 and 6 months, then every 6 months
  Self reported quality of life as measured by the Brief Pain Inventory, European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) C15-PAL, and EORTC QLQ BM22
Progression free survival | up to 3 years
  Progression free survival is defined as time between treatment and first sign of progression of disease
Overall survival | up to 3 years
  Overall survival is defined as time between treatment and death from any cause
Occurrence or progression of vertebral compression fracture (VCF) | up to 12 months
  VCF is defined as new endplate fracture or collapse deformity as compared with before SBRT or EBRT
Occurrence of radiation-induced myelopathy | up to 12 months
  Radiation-induced myelopathy is defined as a diagnosis of exclusion and defined as neurological signs and symptoms consistent with radiation damage in the form of necrosis to the segment of the spinal cord irradiated, without MRI evidence of recurrent or progressive tumour affecting the spinal cord.
Duration of pain relief | at 2, 4, 6, 8 weeks, 3 and 6 months
  Duration of pain relief as measured by the Brief Pain Inventory
Determination of rapidity of pain relief | at 2, 4, 6, 8 weeks, 3 and 6 months
  Rapidity of pain relief as measured by the Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Helena M. Verkooijen, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Pielkenrood BJ, van der Velden JM, van der Linden YM, Bartels MMT, Kasperts N, Verhoeff JJC, Eppinga WSC, Gal R, Verlaan JJ, Verkooijen HML. Pain Response After Stereotactic Body Radiation Therapy Versus Conventional Radiation Therapy in Patients With Bone Metastases-A Phase 2 Randomized Controlled Trial Within a Prospective Cohort. Int J Radiat Oncol Biol Phys. 2021 Jun 1;110(2):358-367. doi: 10.1016/j.ijrobp.2020.11.060. Epub 2020 Dec 14. PMID 33333200
- [Derived] van der Velden JM, Verkooijen HM, Seravalli E, Hes J, Gerlich AS, Kasperts N, Eppinga WS, Verlaan JJ, van Vulpen M. Comparing conVEntional RadioTherapy with stereotactIC body radiotherapy in patients with spinAL metastases: study protocol for an randomized controlled trial following the cohort multiple randomized controlled trial design. BMC Cancer. 2016 Nov 21;16(1):909. doi: 10.1186/s12885-016-2947-0. PMID 27871280
- See also: Related Info — http://www.radiotherapie.nl/